CLINICAL TRIAL: NCT05788458
Title: Effect of Bupivacaine Concentration on Ultrasound Guided Pericapsular Group Nerve Block Efficacy in Hip Surgery Patients: A Randomized Controlled Double Blinded Trial
Brief Title: Effect of Bupivacaine Concentration on Ultrasound Guided Pericapsular Group Nerve Block Efficacy in Hip Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 1-3-2023
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Perioperative Pain
Keywords: pain; positioning; PENG block
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): will receive 20 ml of 0.25 % bupivacaine
  Interventions: Drug: Bupivacain
- Group B (Active Comparator): will receive 20 ml of 0.375 % bupivacaine.
  Interventions: Drug: Bupivacain
- Group C (Active Comparator): will receive 20 ml of 0.5 % bupivacaine.
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — The blocks will be performed in supine position under complete aseptic condition. The site to be blocked will be painted with 5% povidone iodine followed by 70% ethyl alcohol and draped. Linear high-frequency ultrasound probe (7 -15 mhz) (General Electric; GE, "LOGIQ E") will be initially placed in a transverse plane over the anterior superior iliac spine (ASIS) and then alignes to identify the following landmarks: Anterior inferior iliac spine, ilio-pubic eminence, iliopsoas muscle and tendon, the femoral artery, and Pectineus muscle. Point of injection will be musculo-fascial plane between the psoas tendon and ilio-pubic eminence.

SUMMARY:
Fractures in and around the hip are quite common irrespective of both the young and elderly population groups and are associated with extreme pain.The anterior hip capsule is innervated by articular branches of femoral nerve, obturator nerve and accessory obturator nerve (AON) as reported by previous anatomic studies, suggesting that these nerves should be the main targets for hip analgesia, which can be blocked by Peri-capsular nerve group (PENG).

DETAILED DESCRIPTION:
Fractures in and around the hip are quite common irrespective of both the young and elderly population groups and are associated with extreme pain. A hip fracture is a serious injury, with complications that can be life-threatening and is a common orthopedic emergency in the elderly. Early surgery within 48 h of fracture has shown to decrease the complication and mortality rates.

Spinal anaesthesia is the most common mode of anaesthesia used to fix these fractures. Extreme pain due to fracture does not allow ideal positioning for these procedures. and hence a problem to access the subarachnoid space. Inadequate postoperative analgesia can restrict the limb mobility thereby delaying recovery along with increased consumption of opioids.

Effective perioperative analgesia that reduces the requirement of opioids and its adverse effects is essential in this population.

The anterior hip capsule is innervated by articular branches of femoral nerve, obturator nerve and accessory obturator nerve (AON) as reported by previous anatomic studies, suggesting that these nerves should be the main targets for hip analgesia, which can be blocked by Peri-capsular nerve group (PENG) .

PNB with lower volume and higher concentration of local anesthetic was more efficacious than higher volumes and lower concentrations of local anesthetic of equivalent dose.

Using this information, the investigators will conduct this study to evaluate the efficacy of bupivacaine at three different concentration and doses in equivalent volume used in ultrasound guided PENG block for positioning & post-operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* (ASA )classes I and II
* patients of either sex
* above the age of 18 who will undergo hip surgeries( (Dynamic hip screw fixation or hemiarthroplasty)(not older than 2 weeks) with persistent pain and scheduled for surgery under SA with an expected duration of 2.5 hours).

Exclusion Criteria:

* patient's refusal to participate
* any contraindications to SA or peripheral nerve blocks
* history of ischemic heart disease
* patients on opioids for chronic pain
* patients with significant cognitive impairment.
* Patients who have surgery on the hip or spine within 3 months or have no pain while sitting by themselves (resting pain less than 4 on NRS) for SA without any support

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
NRS at rest and on passive 15° limb lifting, EOSP. | 30 minutes after the block
  From 0 to 10 (0 no pain , 10 very sever pain)

SECONDARY OUTCOMES:
NRS over 24 hours | 2,4,8,16,24 hours postoperative
  From 0 to 10 (0 no pain , 10 very sever pain)
Amount of morphine intake. | 24 hours postoperative
  Amount of morphine taken during 24 hours
Quality of recovery score (QoR-15) | at 24 hours postoperative
  This questionnaire covers a total of 15 questions under five clinical dimensions of health; physical comfort (five-item), emotional status (four-item), psychological support (two-item), physical independence (two-item) and pain (twoitem).
  a numerical rating scale of 11 point for each question leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ah Abdelfatah, MD, Principal Investigator — banha faculity of medicine
Locations (1):
- Banha Faculity of Medicine, Banhā, Elqalyoubea, Egypt

REFERENCES:
- [Derived] Abdelfatah FA, Elhadad MA. Effect of bupivacaine concentration on ultrasound-guided pericapsular group nerve block efficacy in hip surgery patients: comparative, randomized, double-blinded clinical trial. Br J Pain. 2024 Oct;18(5):425-432. doi: 10.1177/20494637241262516. Epub 2024 Jun 14. PMID 39355572